CLINICAL TRIAL: NCT05516680
Title: Effects and Central Mechanism of Electroacupuncture and MRI-navigated rTMS for PSD: a fMRI-based Single-center, Randomized, Controlled, Assessor-blinded Trial
Brief Title: Effects and Central Mechanism of Electroacupuncture and MRI-navigated rTMS for PSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-LCYJ-PY-08
Record Dates: First submitted 2022-08-15; First posted 2022-08-25 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-08

CONDITIONS: Post-stroke Depression; Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): electro-acupuncture and MRI-navigated rTMS
  Interventions: Device: electro-acupuncture; Device: MRI-navigated rTMS
- Control group (Active Comparator): MRI-navigated rTMS
  Interventions: Device: MRI-navigated rTMS

INTERVENTIONS:
Device: electro-acupuncture — Acupoints consist of Neiguan (PC6, bilateral), Shuigou (GV26), Sanyinjiao (SP6, affected side), Yintang (EX-HN3), Shangxing (GV23), Baihui (GV20), and Sishencong (EX-HN1). Disposable stainless-steel needles (0.25mm× 40 mm）will be used. After skin disinfection, the acupuncturists will twist and thrust the needle handles to achieve the sensation of achiness, heaviness, and numbness (known as de qi) at all acupoints. Following needle manipulations, electroacupuncture instruments(SDZ-V) will be used to attached the needle handles at EX-HN3, GV23, GV20 and EX-HN1 with a dilatational wave of 5 ~ 10 Hz and a current intensity of 1 ~ 3 mA depending on the patient's tolerance. The needles will be removed after 30 minutes except for GV26 without needle retention. Participants will receive 12-20 electroacupuncture sessions over four weeks at a frequency of 3-5 times per week.
  Arms: Experiment group
Device: MRI-navigated rTMS — MRI:All MRI scans were taken to acquire high-resolution T1-weighted anatomical images on the 3T MRI Scanner. Electromyography(EMG):Surface EMG was used to record MEPs from the abductor pollicis brevis for determining RMT of the non-lesioned motor cortex.A single TMS pulse was delivered to the location to identify the RMT,defined as the minimum intensity capable of evoking at least 5 MEPs of >50 μV in 10 consecutive trials.MRI-navigated rTMS:Using BrainSight system,left DLPFC targeting was individualized by reconstructing MRI data into a 3-dimensional brain image for neuro-navigation. Left DLPFC localization was central middle frontal gyrus,between superior frontal sulcus and middle frontal sulcus based on T1-weighted anatomical images.Focal rTMS was administered using a Magstim Rapid 2 connected to Y125-round coil that was identical.rTMS was applied at 110% RMT to the left DLPFC.At each session,3000 pulses were applied at 10 Hz with a total of 12-20 rTMS sessions over a 4-week period.

SUMMARY:
Introduction:

Post-stroke depression (PSD) is the most common mental complication after stroke and has a serious impact on functional outcomes and quality of life. Antidepressants are the first-line treatment for PSD, but many reported side effects remain. Clinical research and practice guidelines have shown that electro-acupuncture and rTMS have a positive effect on PSD. This trial aims to study the efficacy and safety of electro-acupuncture and a modern MRI-navigated rTMS for PSD and to explore its fMRI-based central mechanism on depression. It is hypothesized that electro-acupuncture and MRI-navigated rTMS treatment improves depressive symptoms, neuro-patho-physiological behaviors, quality of life and central response in PSD.

Methods:

In this randomized, controlled, assessors-blinded trial, sixty-four patients with PSD will be randomly allocated into the experiment group (n=32) or control group(n=32) . The experiment group will receive electro-acupuncture and MRI-navigated rTMS, and the control group will receive MRI-navigated rTMS treatment, in 12-20 sessions over 4 weeks. In addition, ten healthy people for fMRI scanning will be recruited as a healthy control group without any intervention. The primary outcome is the change from baseline in the Hamilton Depression Scale-24 items (HAMD-24) scores at week 4. The primary analysis of central mechanism mainly involves cortical morphology, local spontaneous brain activity, and default mode network (DMN) functional connectivity based on fMRI at 0-wk and 4-wk. Secondary outcomes include the neuro-patho-physiological and quality of life changes in cortical excitability with motor evoked potential test(MEP), National Institutes of Health Stroke Scale(NIHSS), EuroQol Five Dimensions Questionnaire(EQ-5D) Scale, Modified Barthel Index(MBI) Scale and Short Form-Health Scale of Traditional Chinese Medicine(SF-HSTCM). Additional indicators include the Acceptability Questionnaire and Health Economics Evaluation (cost-effectiveness analysis) to assess acceptability and economic practicality of the treatment in study. Outcomes are assessed at baseline and post intervention.

Discussion:

Electro-acupuncture and MRI-navigated rTMS therapy could become an alternative treatment for PSD, and it is expected that this trial will provide reliable clinical evidence and potential effect mechanism for the future use of electro-acupuncture and MRI-navigated rTMS for PSD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients:

* Meet the TCM and Western medicine diagnostic criteria for first onset stroke within 6 months;
* Aged 40-75 years;
* Right-handed;
* Single infarct in basal ganglia (volume:3-5cm);
* Motor evoked potential (MEP) could be recorded by bilateral primary motor cortex (M1) stimulating.
* National Institutes of Health Stroke Scale (NIHSS) score <6;
* Hamilton Depression Scale-24 items (HAMD-24) score > 8;
* Clear consciousness, no hearing and visual impairment, and cooperative physical examination (Glasgow Coma Scale (GCS) score > 8);
* Complete the screening, and sign the informed consent form voluntarily.

Inclusion criteria for healthy subjects:

* Healthy subjects, aged 40-75 years;
* Right-handed;
* HAMD-24 score < 8;
* Sign the informed consent voluntarily.

Exclusion Criteria:

Exclusion criteria for patients:

* Have received other antidepressant therapy or involved in other clinical trials in 2 weeks;
* Infarct was located in the left DLPFC;
* With positive psychiatric history and major trauma exposure history, such as depression, epilepsy, etc. in the past;
* With other serious concomitant diseases (aphasia, severe edema, venous thrombosis, arteriosclerosis occlusion, diabetic vascular disease, peripheral neuropathy, spinal lesions, brain trauma, intracranial infection, brain tumors, etc.), and secondary diseases (heart, liver, renal failure, etc.);
* Infection around acupoints and/or intolerance of acupuncture manipulation;
* With MRI or rTMS contraindications (claustrophobia, metal implants, cochlear implants, impulsator, etc.).

Exclusion criteria for healthy subjects:

* Have involved in other clinical trials in 2 weeks;
* With positive psychiatric history and major trauma exposure history, including depression, epilepsy, etc. in the past;
* With MRI or rTMS contraindications (claustrophobia, metal implants, cochlear implants, impulsator, etc.).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale-24 items scores | change from baseline to week 4
  Reduction rate
fMRI scan | 0 week
  Cortical morphology, local spontaneous brain activity, and default mode network (DMN) functional connectivity
fMRI scan | 4 weeks
  Cortical morphology, local spontaneous brain activity, and default mode network (DMN) functional connectivity

SECONDARY OUTCOMES:
motor evoked potential test | 0 week
  Cortical excitability
motor evoked potential test | 4 weeks
  Cortical excitability
National Institutes of Health Stroke Scale | 0 week
  The minimum and maximum values are 0 and 42 points, and higher scores mean a worse outcome.
National Institutes of Health Stroke Scale | 4 weeks
  The minimum and maximum values are 0 and 42 points, and higher scores mean a worse outcome.
EuroQol Five Dimensions Questionnaire Scale | 0 week
  The minimum and maximum values of utility index are -0.391 and 1 points, and higher scores mean a better outcome.
EuroQol Five Dimensions Questionnaire Scale | 4 weeks
  The minimum and maximum values of utility index are -0.391 and 1 points, and higher scores mean a better outcome.
Modified Barthel Index Scale | 0 week
  The minimum and maximum values are 0 and 100 points, and higher scores mean a better outcome.
Modified Barthel Index Scale | 4 weeks
  The minimum and maximum values are 0 and 100 points, and higher scores mean a better outcome.
Short Form-Health Scale of Traditional Chinese Medicine | 0 week
  The minimum and maximum values are 0 and 130 points, and higher scores mean a worse outcome.
Short Form-Health Scale of Traditional Chinese Medicine | 4 weeks
  The minimum and maximum values are 0 and 130 points, and higher scores mean a worse outcome.

OTHER OUTCOMES:
Acceptability Questionnaire | 4 weeks
  It is involved three levels: "fully accepted", "acceptable" and "not acceptable". The acceptance rate is calculated by the number of "fully accepted" and "acceptable" subjects. And higher rate mean a better outcome.
Health Economics Evaluation | 4 weeks
  Cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be made during the 6 months after the end of study, and the original data can be obtained from the PI if necessary.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the 6 months after the end of study.

REFERENCES:
- [Derived] Lu H, Wang Y, Shen D, Ruan J, Lu J, Wang L, Song Y, Fan J, Li D, Shi L, Xia M, Xu T. Effects and central mechanism of electroacupuncture and MRI-navigated rTMS for PSD: study protocol for an fMRI-based single-center, randomized, controlled, open-label trial. Front Psychiatry. 2024 Jan 4;14:1226777. doi: 10.3389/fpsyt.2023.1226777. eCollection 2023. PMID 38250275